CLINICAL TRIAL: NCT02785666
Title: A Phase III, Multi-center, Open-label Trial to Investigate the Impact of a Treat, Counsel and Cure Strategy in Men Who Have Sex With Men With Hepatitis C Infection in the Swiss HIV Cohort Study
Brief Title: Swiss HCVree Trial
Acronym: HCVree
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BASEC 2016-00131
Record Dates: First submitted 2016-05-17; First posted 2016-05-30 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Hepatitis C; HIV
Keywords: Men who have sex with men; Elimination
MeSH Terms: conditions — Hepatitis C; Homosexuality | interventions — grazoprevir; elbasvir; Ribavirin; elbasvir-grazoprevir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment and behavioural intervention: (Experimental): Treatment intervention: Patients with a replicating GT 1 and/or 4 HCV infection without or with cirrhosis will be treated with grazoprevir/elbasvir (100mg/50mg) for 12 weeks. GT 1a infected patients with baseline RAV's and GT 4 infected patients with a history of prior HCV treatment failure without or with cirrhosis will be treated with the same regimen for 16 weeks, in combination with weight-adjusted ribavirin.
  Behavioural Intervention: Participants with inconsistent condom use with occasional partners will receive the behavioral Intervention and in addition standard of care written and oral information on prevention of HCV reinfection. Study participants with consistent condom use or those reporting inconsistent condom use with occasional partners but not willing to participate in the intervention will receive standard of care written and oral information on prevention of HCV reinfection only
  Interventions: Drug: grazoprevir/elbasvir, ribavirin; Behavioral: Behavioural Intervention

INTERVENTIONS:
Drug: grazoprevir/elbasvir, ribavirin — To investigate the virological efficacy and safety of grazoprevir/elbasvir ±ribavirin for HIV/HCV-coinfected MSM with a GT 1 and/or 4 infection
  Other Names: Zepatier, Rebetol
Behavioral: Behavioural Intervention — To counsel the targeted population with a behavioral intervention regarding the reduction of sexual risk behaviour and recreational drug use.

SUMMARY:
The investigators aim at investigating the efficacy of grazoprevir/elbasvir ±ribavirin in HIV-positive MSM participating in the SHCS in a broader setting of coinfected MSM. The study pursues a comprehensive approach of a treat, counsel and cure strategy exploring the impact of such a strategy in a representative HIV/HCV-coinfected MSM population. This study is a nested project of the Swiss HIV Cohort Study entitled "The Swiss HCVree Trial".

DETAILED DESCRIPTION:
The prevalence of hepatitis C virus (HCV) infection is increasing in HIV-positive men who have sex with men (MSM) participating in the Swiss HIV Cohort Study (SHCS). MSM with high-risk sexual behaviour are recognized to be the main drivers of the current HCV epidemic. However, in Switzerland treatment with the newest available direct acting agents (DAAs) is currently restricted to patients with a METAVIR fibrosis score ≥2 (i.e., patients with beginning or advanced liver fibrosis or cirrhosis) by the federal office of public health due to the tremendous costs of these DAAs. Within the study population (i.e. HIV-infected MSM with a replicating HCV-infection in Switzerland), about 90% of individuals have a METAVIR fibrosis score <2. As a consequence, HCV therapy with new DAAs is not covered by health insurances for the majority of this population. However, there is evidence that HCV treatment should not be delayed until the development of advanced liver disease. Treating HIV/HCV-coinfected individuals independently of their liver fibrosis score can prevent the development of liver related complications and the transmission of HCV infection.

The once daily oral combination regimen grazoprevir/elbasvir was approved by the Food and Drug Administration (FDA) in January 2016 for the treatment of genotype (GT) 1 and 4 HCV infection in mono- and HIV/HCV coinfected patients. In phase III clinical trial, a 12-week course of grazoprevir/elbasvir showed high efficacy with sustained virologic response (SVR) rates of ≥95%, and favourable tolerability. A 16 weeks treatment with grazoprevir/elbasvir in combination with weight-adjusted ribavirin is necessary in GT 1a infected patients with baseline resistance associated variants (RAV's) and GT 4 infected patients with a history of prior failure to HCV-treatment. Grazoprevir/elbasvir has only robust data from phase 2 and 3 clinical trials for GT 1, 4 HCV infections.

Of note, GT 1, 4 infections account for ~90% of HCV infections in the MSM population in the SHCS.

HCV reinfection remains a concern among MSM, who can be re-exposed to HCV through high-risk sexual behaviours after successful HCV treatment. A recent review shows evidence that behavioural interventions in high risk MSM have the potential to be effective at least in short term reduction of sexual risk behaviours.

To date the knowledge about the HCV-specific immune responses during DAA treatment is sparse. An effective adaptive cellular immunity is known to play a crucial role in spontaneous viral eradication after primary infection.

The investigators aim at investigating the efficacy of grazoprevir/elbasvir ±ribavirin in HIV-positive MSM participating in the SHCS in a broader setting of coinfected MSM. The study pursues a comprehensive approach of a treat, counsel and cure strategy exploring the impact of such a strategy in a representative HIV/HCV-coinfected MSM population. This study is a nested project of the Swiss HIV Cohort Study entitled "The Swiss HCVree Trial".

ELIGIBILITY:
Inclusion Criteria:

* Informed consent documented by signature
* Participation in the SHCS
* Male individual ≥18 years old
* Homosexual or bisexual preference/transmission mode according to the SHCS entry state and/or in the opinion of the study physician.
* Replicating HCV infection (i.e., positive HCV-RNA-test).
* HCV GT 1 and/or 4 infection.

Exclusion Criteria:

* Contraindications to grazoprevir/elbasvir and ribavirin due to significant drug-drug interactions (DDI) (e.g., HIV protease inhibitors) according to the Liverpool drug-interaction data base.
* Contraindications to grazoprevir/elbasvir and ribavirin, e.g. known hypersensitivity or allergy to the class of drugs or the investigational product.
* Participant is under the age of legal consent, is mentally or legally incapacitated, has significant emotional problems at the time of pre-study screening visit or expected during the conduct of the study or has a history of a clinically significant psychiatric disorder which, in the opinion of the investigator, would interfere with the study procedures.
* Inability to follow the study procedures (e.g. language barriers, psychiatric disorders
* Known or suspected non-adherence to study-procedures.
* Currently participating or has participated in a study with an investigational compound within 30 days of signing informed consent and is not willing to refrain from participating in another such study during the course of this study.
* Enrolment of the investigator, his/her family members, employees and other dependent persons.
* Participant suffers from clinically significant concomitant diseases (for the detailed list of diseases we refer to the according section of this protocol).
* Participant has a history of malignancy ≤5 years prior to signing informed consent or is under evaluation for other active or suspected malignancy.
* Participant has a history of opportunistic infection in the preceding 6 months prior to screening.
* Participants with mixed HCV infection of genotype 1, 4 or 6 with genotype 2, 3 or 5.
* Participant is coinfected with HBV-DNA positive hepatitis B virus (of note, HBsAg positive individuals with suppressed HBV-DNA might be included).
* Participant has evidence of decompensated liver disease.
* Liver cirrhosis Child-Pugh Class B or C, or who have a Pugh-Turcotte (CPT) score >5,
* Participant has cirrhosis and liver imaging within 6 months of Day 1 showing evidence of hepatocellular carcinoma (HCC) or is under evaluation for HCC.
* Participant has clinically-relevant drug or alcohol abuse at the PI's discretion within 12 months of screening.
* Participant is a male whose female partner(s) is/are pregnant (this is a contraindication for ribavirin use)
* Participant has exclusionary laboratory values at the screening visit (for the table containing these laboratory values we refer to the according section of this protocol).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-06; Primary Completion 2018-04 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Virological efficacy of grazoprevir/elbasvir ±ribavirin: SVR rates at week 12 after treatment stop. | 12 weeks after treatment stopp, i.e. week 24.
  The main analysis will be the evaluation of SVR 12 weeks after end of treatment (SVR12). We will determine the proportion of patients with an SVR12 (HCV viral load< 20 copies per ml) in intention to treat analyses including all patients who have received at least one dose of the study compound. Per protocol analyses will also be performed.

SECONDARY OUTCOMES:
Safety of grazoprevir/elbasvir ±ribavirin: frequency of adverse events and serious adverse events. | At week 0, week 4, week 6, week 8, week 12, week 16, and week 24.
  AE will be assessed at every study-visit using standardized AE forms from the electronic case Report form
Change in condom use before and after the behavioural Intervention | At week 0, week 12, and week 24.
  Changes in condom use will be assessed as mediators for behaviour change. The behavioral intervention will be evaluated as a case-control study with the behavioural intervention as the exposure and a switch from "reporting condom-less sex" to "not reporting condom-less sex" as the outcome.
Change in recreational drug use before and after the behavioural intervention | At week 0, week 12, and week 24.
  Changes in recreational drug use will be assessed as mediators for behaviour change. The behavioral intervention will be evaluated as a case-control study with the behavioural intervention as the exposure and a switch from "reporting recreational drug use" to "not reporting recreational drug use" as the outcome.
Change in condom use attitude before and after the behavioural intervention | At week 0, week 12, and week 24.
  Changes in attitude of condom use use will be assessed as mediators for behaviour change. The behavioral intervention will be evaluated as a case-control study with the behavioural intervention as the exposure and a switch from "reporting condom-less sex" to "not reporting condom-less sex" as the outcom
Change in condom use self-efficacy before and after the behavioural intervention | At week 0, week 12, and week 24.
  Changes in attitude of condom use self-efficacy will be assessed as mediators for behaviour change. The behavioral intervention will be evaluated as a case-control study with the behavioural intervention as the exposure and a switch from "reporting condom-less sex" to "not reporting condom-less sex" as the outcom
Change in condom use behaviour before and after the behavioural intervention | At week 0, week 12, and week 24.
  Changes in attitude of condom use will be assessed as mediators for behaviour change. The behavioral intervention will be evaluated as a case-control study with the behavioural intervention as the exposure and a switch from "reporting condom-less sex" to "not reporting condom-less sex" as the outcom
Change in recreational drug use attitude before and after the behavioural intervention | At week 0, week 12, and week 24.
  Changes in recreational drug use attitude will be assessed as mediators for behaviour change. The behavioral intervention will be evaluated as a case-control study with the behavioural intervention as the exposure and a switch from "reporting recreational drug use" to "not reporting recreational drug use" as the outcome.
Change in recreational drug use behaviour before and after the behavioural intervention | At week 0, week 12, and week 24.
  Changes in recreational drug use behaviour will be assessed as mediators for behaviour change. The behavioral intervention will be evaluated as a case-control study with the behavioural intervention as the exposure and a switch from "reporting recreational drug use" to "not reporting recreational drug use" as the outcome.
Change in recreational drug use self-efficacy before and after the behavioural intervention | At week 0, week 12, and week 24.
  Changes in recreational drug use self-efficacy will be assessed as mediators for behaviour change. The behavioral intervention will be evaluated as a case-control study with the behavioural intervention as the exposure and a switch from "reporting recreational drug use" to "not reporting recreational drug use" as the outcome.
HCV treatment uptake: proportion of potentially eligible MSM participating in this study. | At week 0
  Treatment uptake will be compared according to demographical and clinical characteristics. Descriptive statistics will be used to assess risk factors for not initiating HCV therapy.
Identification of presumed places of HCV acquisition and modes of HCV transmission: evaluation of patient's questionnaires | At week 0
  All patients will fill out an patient questionnaire at visit 1 where they are asked to provide information on the potential transmission mode (e.g., unprotected anal intercourse, intravenous drug use) of the HCV infection and the presumed places of acquisition (e.g. foreign country, Switzerland, city). This questionnairs will be analysed qualitatively.
Barriers to treatment: systematic documentation of exclusion reasons for HCV treatment by patient's questionnaire | At week 0
  Reasons not to start HCV treatment will be compared according to demographical and clinical characteristics. Descriptive statistics will be used to assess risk factors for not initiating HCV therapy.
Adherence to HCV treatment: proportion of patients which are adherent to ≥95% of prescribed pills | At week 0, week 4, week 6, week 8, week 12, and week 24.
  Adherence will be defined as the proportion of study drug doses taken. Acceptable adherence will be met if at least 95% of the prescribed tablets are taken. Predictors of non-adherence will be assessed using logistic regression and adherence will be included as an explanatory variable into the model evaluating predictors of the primary outcome.
Impact of resistance associated variants: SVR 12 in GT 1a infected individuals stratified by presence of baseline RAV's. | At week 24, i.e. 12 weeks after treament stopp
  In every patient with a GT 1a HCV infection a HCV resistance test will pe performed to determine resistance associated variants (RAV's) at baseline. Based on the presence of baseline RAVs the treatment duration will be prolonged to 16 weeks in addition to ribavirin as add-on to grazoprevir/elbasvir. The SVR 12 rates will then be analysed comparing the patients with and without baseline RAVs.
Assessment of HCV-specific cellular immune response: changes of HCV-specific T-cell functionality by ex vivo fluorescence-activated cell sorting (FACS) before and after DAA therapy | At week 0, and week 24
  For the assessment of the cellular immune responses descriptive statistics will be used to compare changes before and after medical intervention and regression analysis to assess the influence of the immune responses on treatment failure and HCV re-infection.
Assessment of HCV-specific cellular immune response: changes of HCV-specific T-cell phenotype by ex vivo fluorescence-activated cell sorting (FACS) before and after DAA therapy | At week 0, and week 24
  For the assessment of the cellular immune responses descriptive statistics will be used to compare changes before and after medical intervention and regression analysis to assess the influence of the immune responses on treatment failure and HCV re-infection.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique L Braun, MD, Principal Investigator — University Hospital Zurich, University of Zurich
Locations (1):
- Division of Infectious Diseases and Hospital Epidemiology, University Hospital Zurich, University of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kusejko K, Salazar-Vizcaya L, Shah C, Stockle M, Beguelin C, Schmid P, Ongaro M, Darling K, Bernasconi E, Rauch A, Kouyos RD, Gunthard HF, Boni J, Fehr JS, Braun DL; Swiss HIV Cohort Study. Sustained Effect on Hepatitis C Elimination Among Men Who Have Sex With Men in the Swiss HIV Cohort Study: A Systematic Re-Screening for Hepatitis C RNA Two Years Following a Nation-Wide Elimination Program. Clin Infect Dis. 2022 Nov 14;75(10):1723-1731. doi: 10.1093/cid/ciac273. PMID 35404384
- [Derived] Kunzler-Heule P, Fierz K, Schmidt AJ, Rasi M, Bogdanovic J, Kocher A, Engberg S, Battegay M, Nostlinger C, Lehner A, Kouyos R, Schmid P, Braun DL, Fehr J, Nicca D. Response to a sexual risk reduction intervention provided in combination with hepatitis C treatment by HIV/HCV co-infected men who have sex with men: a reflexive thematic analysis. BMC Infect Dis. 2021 Apr 6;21(1):319. doi: 10.1186/s12879-021-06003-z. PMID 33823783
- [Derived] Braun DL, Hampel B, Ledergerber B, Grube C, Nguyen H, Kunzler-Heule P, Shah C, Salazar-Vizcaya L, Conen A, Flepp M, Stockle M, Beguelin C, Schmid P, Rougemont M, Delaloye J, Bernasconi E, Nicca D, Boni J, Rauch A, Kouyos RD, Gunthard HF, Fehr JS. A Treatment-as-Prevention Trial to Eliminate Hepatitis C Among Men Who Have Sex With Men Living With Human Immunodeficiency Virus (HIV) in the Swiss HIV Cohort Study. Clin Infect Dis. 2021 Oct 5;73(7):e2194-e2202. doi: 10.1093/cid/ciaa1124. PMID 32761122
- [Derived] Kunzler-Heule P, Engberg S, Battegay M, Schmidt AJ, Fierz K, Nguyen H, Kocher A, Nostlinger C, Hampel B, Stockle M, Beguelin C, Delaloye J, Schmid P, Flepp M, Rougement M, Braun DL, Fehr J, Nicca D; Swiss HIV Cohort Study (SHCS). Screening HIV-positive men who have sex with men for hepatitis C re-infection risk: is a single question on condom-use enough? A sensitivity analysis. BMC Infect Dis. 2019 Sep 18;19(1):821. doi: 10.1186/s12879-019-4456-7. PMID 31533734
- [Derived] Braun DL, Hampel B, Martin E, Kouyos R, Kusejko K, Grube C, Flepp M, Stockle M, Conen A, Beguelin C, Schmid P, Delaloye J, Rougemont M, Bernasconi E, Rauch A, Gunthard HF, Boni J, Fehr JS; Swiss HIV Cohort Study. High Number of Potential Transmitters Revealed in a Population-based Systematic Hepatitis C Virus RNA Screening Among Human Immunodeficiency Virus-infected Men Who Have Sex With Men. Clin Infect Dis. 2019 Feb 1;68(4):561-568. doi: 10.1093/cid/ciy545. PMID 30107494
- [Derived] Braun DL, Hampel B, Kouyos R, Nguyen H, Shah C, Flepp M, Stockle M, Conen A, Beguelin C, Kunzler-Heule P, Nicca D, Schmid P, Delaloye J, Rougemont M, Bernasconi E, Rauch A, Gunthard HF, Boni J, Fehr JS; Swiss HIV Cohort Study. High Cure Rates With Grazoprevir-Elbasvir With or Without Ribavirin Guided by Genotypic Resistance Testing Among Human Immunodeficiency Virus/Hepatitis C Virus-coinfected Men Who Have Sex With Men. Clin Infect Dis. 2019 Feb 1;68(4):569-576. doi: 10.1093/cid/ciy547. PMID 30107485